CLINICAL TRIAL: NCT06382415
Title: Effect of Organ/Space Surgical Site Infection After Rectal Cancer Resection on Five-year Recurrence and Survival Rates. A Population-based Cohort Study of 2208 Patients
Brief Title: Organ/Space Surgical Site Infection and Recurrence and Survival in Rectal Cancer Surgery
Acronym: VINCat_PDO_2
Status: Completed | Type: Observational
Sponsor: Hospital de Granollers (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other); Institut Català d'Oncologia (Other)
Responsible Party: Principal Investigator, Josep M Badia, Prof, Hospital de Granollers
Other Study IDs: VINCat_PDO_2
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Rectal Cancer; Organ-Space Surgical Site Infection
Keywords: Surgical Site Infection; Rectal cancer; Rectal Surgery; Survival; Recurrence
MeSH Terms: conditions — Rectal Neoplasms; Surgical Wound Infection; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients operated on rectal cancer: Patients operated on rectal cancer, included in two compulsory audits of the Catalan Cancer registry and in the Catalan Infection Surveillance Program, who suffered an organ-space surgical infection.

SUMMARY:
In rectal cancer surgery, the organ/space surgical site infection (O/S-SSI) has an impact on patient's prognosis. Its influence in the oncologic outcomes remains controversial. The main objective is to assess the possible effect of O/S-SSI on long-term overall survival and cancer recurrence.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common malignancy worldwide and the fourth leading cause of cancer death in both sexes, accounting for 30-35% of all tumours originating in the rectum. Although the introduction of total mesorectal excision and the use of neoadjuvant chemoradiation have improved the oncological outcome in patients with rectal cancer operated with curative intent, the 5-year recurrence rate remains around 20%, with tumour stage being the most important prognostic factor. Other tumour-related factors, such as lymphovascular, perineural and extramural vascular invasion, as well as response to neoadjuvant treatment, have also been shown to be reliable predictors of recurrence. However, surgery-related factors, such as the quality of surgical resection as well as the occurrence of postoperative complications, may have a profound impact on these outcomes.

Anastomotic leakage is one of the most serious complications of colorectal surgery and its frequency ranges from 3 to 21% depending on the location of the tumour and the definition of anastomotic leakage used. This complication is associated with considerable morbidity and mortality and may affect quality of life. Several studies have shown that anastomotic leakage and subsequent organ-space infection (O/S-SSI) are also associated with higher rates of tumour recurrence and cancer-specific mortality. A recent meta-analysis involving 43 studies with a total of 154,981 patients undergoing colorectal cancer surgery found that postoperative O/S-SSI and anastomotic leakage had a significant negative impact on disease-free survival, local recurrence and overall recurrence. This association has also been reported after resection of liver metastases and other gastrointestinal malignancies. In addition, the severity of postoperative infection has also been correlated with increased risk of recurrence.

However, these results have not been confirmed in other studies. In our setting, the development of anastomotic leaks did not affect the risk of local recurrence, overall recurrence, overall survival or cancer-specific survival in a multicentre observational study using prospectively collected data from 1181 consecutive rectal cancer patients in 22 hospitals included in the Spanish Rectal Cancer Project. These results were consistent with data reported by national colorectal cancer registries such as those of Denmark and Sweden, among others. Therefore, the question of whether anastomotic leakage contributes to disease recurrence remains controversial and requires further research.

In an attempt to clarify this controversy, a population-based study was conducted to assess the influence of O/S-SSI on recurrence and survival outcomes in patients who had undergone curative surgery for rectal cancer in hospitals integrated in the Public Health System of Catalonia (Spain) at 5-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Eligible patients with tumour ≤ 13 cm from anal verge, as measured by Magnetic Resonance Imaging
* Primary adenocarcinoma
* Oncological resection with curative intent
* Cancer stages: I-II-III

Exclusion Criteria:

* Transanal local resection
* Emergency colorectal surgeries
* Presence of metastases found in the diagnostic process or during the surgical procedure
* Recurrence of the disease treated before the study period
* Non-resectable tumour or palliative surgery
* Patients operated in private centres

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated on rectal surgery for rectal cancer in Catalonia, Spain.
Sampling Method: Non-Probability Sample
Enrollment: 3826 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of overall cancer recurrence | 5 years (from date of the surgical procedure until 5 years post-surgery)
  Overall cancer recurrence included locoregional recurrence and systemic recurrence. Locoregional recurrence was defined as tumor linked with surgical site (anastomosis, tumor bed or mesentery), and systemic recurrence as the disease spreading to organs outside the surgical field, such as the liver, lungs, bones, or brain, confirmed histologically or by imaging.
Overall survival | From date of the surgical procedure until the date of death, assessed up to 5 years
  Overall survival (OS) was defined as the time from surgery to death by any cause.

SECONDARY OUTCOMES:
Rate of Organ-space surgical site infection | 30 days
  As described by the Centers for Disease Control: an infection occurring within 30 days of the surgical procedure and involves any part of the body deeper than the fascial/muscle layers that is opened or manipulated during surgery. In addition, the patient must present at least one of the following associated events: a purulent drainage from a drain placed into the organ/space
Rate of surgical complications | 30 days
  Postoperative complications were classified in accordance with the Clavien-Dindo Classification

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Català d'Oncologia, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Restrictions apply to the availability of these data, which belong to two national databases and are not publicly available. Data was obtained from the Catalan Cancer Plan and VINCat, and are only available with the permission of their Technical Committees.